CLINICAL TRIAL: NCT02763735
Title: Metabolic Intervention in the Right Ventricle in Pulmonary Arterial Hypertension
Brief Title: Right Ventricular Metabolism in Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Evan Brittain, Assistant Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 131271
Record Dates: First submitted 2016-04-28; First posted 2016-05-05 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Arterial Hypertension; Healthy
Keywords: Pulmonary arterial hypertension; Right ventricle; Right ventricular function; Metabolism; Non-invasive imaging; Healthy Subjects
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pulmonary Arterial Hypertension: Patients diagnosed with idiopathic or heritable pulmonary arterial hypertension according to consensus guidelines. RV oxidative metabolism and glycolysis will be measured using PET 11C acetate and [18F]fluoro-deoxy-Dglucose (FDG) imaging and measure myocardial lipid accumulation using MRS imaging.
- Subjects without cardiopulmonary disease: Subjects without known cardiopulmonary disease. RV oxidative metabolism and glycolysis will be measured using PET 11C acetate and [18F]fluoro-deoxy-Dglucose (FDG) imaging and measure myocardial lipid accumulation using MRS imaging

SUMMARY:
The purpose of this study is to use non-invasive imaging to determine the metabolic phenotype of the right ventricle in patients with pulmonary arterial hypertension across a spectrum of disease severity.

DETAILED DESCRIPTION:
Current medical therapy for pulmonary arterial hypertension (PAH) is aimed at reducing pulmonary vascular resistance (PVR) but not ameliorating right ventricular (RV) failure, the major cause of death. There are no RV-specific therapies currently available for PAH, in part because the pathophysiology of RV failure is poorly understood.

The investigators hypothesize that the RV in PAH develops a distinct metabolic pattern characterized by increased glycolysis, impaired oxidative metabolism and lipid deposition, which are associated with RV failure.

Specific Aim 1. To test the hypothesis that the RV in human PAH exhibits lipid deposition, increased glycolysis and impaired fatty acid oxidation. The investigators will measure RV oxidative metabolism and glycolysis in PAH patients and controls using positron emission tomography 11C acetate and [18F]fluoro-deoxy-D-glucose imaging and measure myocardial lipid accumulation using magnetic resonance spectroscopy imaging.

Specific Aim 2. To test the hypothesis that an abnormal RV metabolic profile is associated with RV dysfunction and reduced exercise capacity in PAH. PET and MRS findings will be correlated with RV function, patient exercise capacity and a blood metabolic profile.

ELIGIBILITY:
Inclusion Criteria:

* Heritable or idiopathic PAH
* 18 years or older
* Able to give informed consent

Exclusion Criteria:

* Pregnancy
* Type 1 diabetes mellitus
* Prednisone use
* PAH associated with any condition other than idiopathic or heritable
* Implanted ferromagnetic material incompatible with MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pulmonary Arterial Hypertension (heritable or idiopathic) Healthy Subjects
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-06; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Right ventricular oxygen consumption divided by the rate pressure product | At time of C11 acetate PET scan
  kmono divided by the rate pressure product (heart rate X systolic blood pressure)

SECONDARY OUTCOMES:
Right ventricular oxygen consumption (kmono) | At time of C11 acetate PET scan
Right ventricular glucose uptake (standardized uptake value) | At time of 18-FDG PET scan
Percent myocardial triglyceride content | At time of cardiac magnetic resonance imaging
  Percent of myocardial triglyceride measured in the interventricular septum
Correlation of kmono, kmono/RPP, FDG uptake, and myocardial triglyceride content with right ventricular function | Day 1
Correlation of kmono, kmono/RPP, FDG uptake, and myocardial triglyceride content with six minute walk distance | Day 1
Correlation of kmono, kmono/RPP, FDG uptake, and myocardial triglyceride content with plasma metabolic profile | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No